CLINICAL TRIAL: NCT00561938
Title: Confocal Laser Endomicroscopy in the Digestive Tract: A Multicentre French Pilot Study.
Brief Title: Confocal Laser Endomicroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BRD 07/3-Q
Record Dates: First submitted 2007-11-20; First posted 2007-11-21 (Estimated); Last update posted 2009-02-25 (Estimated); Status verified 2009-02

CONDITIONS: Digestive System Diseases
Keywords: Confocal laser endomicroscopy; cancerous and non-cancerous conditions; tolerance; intravenous fluorescein; Digestive symptoms or disease requiring an endoscopy procedure (upper GI endoscopy or colonoscopy) performed under general anaesthesia
MeSH Terms: conditions — Digestive System Diseases | interventions — Colonoscopy; Endoscopy

INTERVENTIONS:
Procedure: Colonoscopy — microscope with a confocal window in its distal part. During ongoing endoscopy, 5 mL of 10% fluorescein (Novartis) will be injected intravenously to perform CLE imaging. In brief, CLE images are obtained few seconds after fluorescein injection by gentle positioning of the confocal window in contact with the digestive mucosa. To stabilize images, some suction can be applied using the operating channel of the endoscope. CLE images ('optical biopsies') will be stored and 1-2 standard biopsies will be performed in the examined area in order to further compare optical and standard biopsies. The overall duration of the procedure will be limited to 1 hour. During and after the procedure, patients will be monitored and surveyed continuously by anaesthesiologist. General tolerance and potential late adverse events will be assessed by the careful inquiry performed 1 month after the procedure by consultant gastroenterologist.
Procedure: Endoscopy — After obtaining a written informed consent from all the patients, standard upper GI endoscopy or colonoscopy will be performed under general anaesthesia using a videoendoscope EC-3870 (Pentax), which includes a miniaturized microscope with a confocal window in its distal part. During ongoing endoscopy, 5 mL of 10% fluorescein (Novartis) will be injected intravenously to perform CLE imaging. In brief, CLE images are obtained few seconds after fluorescein injection by gentle positioning of the confocal window in contact with the digestive mucosa. To stabilize images, some suction can be applied using the operating channel of the endoscope. CLE images ('optical biopsies') will be stored and 1-2 standard biopsies will be performed in the examined area in order to further compare optical and standard biopsies. The overall duration of the procedure will be limited to 1 hour. During and after the procedure, patients will be monitored and surveyed continuously by anaesthesiologist.

SUMMARY:
Confocal laser endomicroscopy (CLE) is a new diagnostic technique that allows microscopic examination of the digestive mucosa during ongoing endoscopy. Different types of tissue and diseases can be diagnosed immediately, and analysis of the in vivo microarchitecture is helpful to better target standard biopsies and reduce the number of biopsies required. CLE necessitates an intravenous injection of a fluorescent marker, e.g. fluorescein, to obtain 'optical biopsies' with a high level of magnification (up to 1000 fold). To date, more than 1000 endomicroscopy procedures have been performed in the world and different publications have shown the safety, feasibility and excellent diagnostic yield of CLE. No complication related to IV injection of fluorescein has been reported. However, all these data come from a very limited number of expert centres and need to be confirmed and validated at the multicenter level. The aims of this multicenter trial are: 1) to standardize CLE in all centres equipped in France, 2) to ensure the safety of intravenous fluorescein injection, 3) to test the diagnostic value of CLE in various conditions representative of the large spectrum of different cancerous and non-cancerous digestive diseases.

ELIGIBILITY:
Inclusion criteria:

* Patient between 18 to 70 years-old
* Symptoms or disease requiring an upper GI endoscopy or a colonoscopy performed under general anaesthesia
* Written informed consent obtained

Exclusion criteria:

* No indication for upper GI endoscopy or colonoscopy
* Treatment by beta-blockers
* Coagulopathy
* Dialysis for impaired renal function
* Pregnancy or breast-feeding
* Known allergy to fluorescein
* Pace-maker
* Severe cardiac or liver disease
* Emergency context- Zenker's diverticulum (for upper GI endoscopy) or recently complicated colonic diverticulosis (for colonoscopy)
* Patient's refusal

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2007-06; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
To establish a safe and standardized practice of CLE in France, which should give a possibility, by providing high quality optical biopsies, to perform in vivo diagnosis of different digestive diseases

SECONDARY OUTCOMES:
To assess the tolerance of CLE in terms of frequency and gravity of potential adverse events related to the injection of fluorescein
To assess the diagnostic yield of CLE in various clinical conditions (cancerous and non-cancerous diseases) by comparing optical biopsies with standard histology
To assess the interobserver agreement for this technique, using a database of optical biopsies created at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Galmiche, PhD, Principal Investigator — Nantes University Hospital
Locations (5):
- France (5):
  - Service d'Hépato-Gastroentérologie, Centre Hospitalier Lyon Sud, Lyon
  - Service d'Hépato-Gastroentérologie, Institut Paoli Calmettes, Marseille
  - Service d'Hépato-Gastroentérologie, CHU Nantes, Nantes
  - Service d' hépato-gastro-entérologie, CHU de ROUEN, Rouen
  - CHU de Rangueil, Toulouse